CLINICAL TRIAL: NCT01979848
Title: MRI (Magnetic Resonance Imaging) Temperature Mapping of the Prostate and Urogenital Pelvis Cooled by an Endorectal Balloon
Brief Title: MRI Temperature Mapping of the Prostate and Urogenital Pelvis Cooled by an Endorectal Balloon
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Thomas E. Ahlering, Vice Chairman and Urology Professor, University of California, Irvine
Other Study IDs: 2012-8932; UCI 12-25 (Other: University of California Irvine)
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Prostate Cancer; Hypothermia; Urinary Incontinence; Erectile Dysfunction
Keywords: continence outcomes; sexual function; Robotic Assisted Radical Prostatectomy; thermal imaging; localized hypothermia
MeSH Terms: conditions — Prostatic Neoplasms; Hypothermia; Urinary Incontinence; Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MRI Mapping Group: After Subjects arrive at the MRI facility, subjects will fill out a medical questionnaire that will be used to determine whether a MRI study can be performed. The investigators will determine whether there are any problems that make the subject not suitable for participating in this study.

SUMMARY:
Urinary incontinence and sexual dysfunction are potential side effects for men undergoing the successful removal of the cancerous prostate via surgery. Hypothermic cooling via the investigational Endorectal Cooling Balloon has been shown by our group to significantly reduce long term urinary incontinence and may reduce sexual dysfunction in men after robotic prostatectomy, and improve the patient's long term quality of life (QOL). However before successful translation of the endorectal balloon can proceed into the world wide usage, we must understand:

1. How effectively the tissues for continence and sexual function are cooled within the pelvis.
2. What is the capacity of vascularized structures (i.e. the neurovascular bundle) to 'cool sink' or diminish the effective cooling and
3. Determine if the endorectal balloon can be re-designed for improved QOL outcomes in men.

This research study marries two new techniques of Thermal MRI imaging and Endorectal cooling for prostate cancer surgery. MRI is non-invasive. A simple confirmation of effective hypothermic cooling can be achieved by novel MRI thermal mapping of the cooling gradient as it comprehensively sweeps through the rectum across the urogenital pelvis. MRI with temperature adaptive software can accurately map these gradients with non-invasive technique, and answer formidable questions of the effectiveness of hypothermic cooling of the prostate and its direct translation into improved continence and sexual function after surgery. The purpose of this research study is to use Magnetic Resonance Imaging (MRI) and Thermal MRI with subjects who will receive the investigational endorectal cooling balloon to help further understand how the cooling balloon works, which may translate to other uses in the future, including the diagnosis of patients at a high risk of developing prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer is the second most frequent cause of cancer death in men and it accounts for 11% of all male cancers. Radical prostatectomy remains the gold standard for localized disease, offering the advantage of precise staging and grading and the real possibility of disease eradication. In the US there are approximately 100,000 radical prostatectomies (RP) performed for prostate cancer annually. However, there are two major challenges to the quality of life outcomes after radical prostatectomy: preserving urinary continence, and sexual function. The quality of life (QOL) after radical prostatectomy relies on the return of continence and sexual function after surgery to their pre-operative 'normal' status. The main factor which determines potency rates for patients is whether or not the nerves at the Neurovascular Bundles (NVB), are spared, and it may take years for sexual function to return. This may be due to the nerve injury from the nerve trauma in the surgical procedure. Similarly, a major factor involved in post-radical prostatectomy incontinence is preservation of the nerves that control the external urethral sphincter, bladder, and urogenital diaphragm. Also Inflammation from surgical removal of the prostate not only affects nerves, but also may directly damage the bladder, urethra, and pelvic floor. Effective strategies to prevent this damage are currently lacking. One stratagem to prevent or minimize such damage, is the use of local hypothermia with ice or cold irrigation around the nerves and tissues prior to, during, and after the injury has occurred. In numerous experimental models of central and peripheral nervous system injury, the use of moderate hypothermia (i.e. 28-33oC) has been shown to provide dramatic neuroprotection safely in humans, during cardiac, kidney, and brain surgery for many years.

ELIGIBILITY:
Inclusion Criteria:

1. A male older than 21 years of age and under age of 80 who does not have prostate cancer and is not enrolled in UCI HS# 2008-6397 (2 male adults to test the MR Temperature Mapping calibration).

   a. CONTROLS: Option for two non-cancer adult male volunteers > 21 years old, to test MR Temperature Mapping calibration. These men are not scheduled for / will not undergo the prostatectomy and related thermometry MRI.
2. A male older than 40 years of age who has confirmed prostate cancer and has decided to receive prostatectomy; and have enrolled in UCI HS# 2008-6397 or will be receiving the Endorectal Cooling balloon outside of UCI HS# 2008-6397 as part of a compassionate use.

Exclusion Criteria:

1. Have implanted prosthetic heart valves, pacemaker, neuro-stimulation devices, surgical clips (hemostatic clips) or other metallic implants,
2. Have engaged in occupations or activities which may cause accidental lodging of ferromagnetic materials, or have imbedded metal fragments from military activities,
3. Have a history of renal disease and determined by the doctor not suitable for receiving injection of MR contrast agent,
4. Unable to lie down still for 60 minutes.
5. Woman or minor

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male volunteers (n=2) to test the MR Temperature Mapping calibration
  AND
  Men who will be undergoing robotic assisted radical prostatectomy will undergo the thermal MRI scans
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Describe cooling based on MRI thermal mapping in terms a) change in temperature over time at 5 locations and by b) thermal map of tissue volume at various time points | One session MRI thermal mapping
  During pre and post hypothermia, initial temperatures will be measured simultaneously on five 3-mm-thick image slices that covered the target. The thermometry scan can be repeated every 6 s. Tissue temperature map is measured by magnetic resonance thermometry (echo planar imaging with multiphase; field of view: 25 × 25 cm; matrix 256 × 256; number of excitations: 1; repetition time: 545 ms; echo time: 20 ms; flip angle: 20°; slice thickness: 3 mm); (b) a thermal map of the tissue volume will be superimposed on the anatomical image.

SECONDARY OUTCOMES:
Describe associations between temperature (at 5 locations) and time to continence. | 30 days and 60 days after Robotic surgery
  Before the subject's scheduled radical prostatectomy surgery, they will have an MRI combined with an cooling endorectal balloon (this study), which will 1. Show the dimensions of their lower pelvis, including the prostate, and 2.Measure how cold the tissue around the prostate becomes using the cooling balloon. The thermal MRI images will allow elucidation of temperatures at specified anatomic locations and their changes over time. Data will be described using means for normally distributed continuous variables. We will test for associations between temperature and continence using t-tests to compare temperature change between those who achieve continence at 30 and 60 days and those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Ahlering, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Background] Finley DS, Osann K, Skarecky D, Ahlering TE. Hypothermic nerve-sparing radical prostatectomy: rationale, feasibility, and effect on early continence. Urology. 2009 Apr;73(4):691-6. doi: 10.1016/j.urology.2008.09.085. Epub 2009 Feb 28. PMID 19250660
- [Background] Finley DS, Osann K, Chang A, Santos R, Skarecky D, Ahlering TE. Hypothermic robotic radical prostatectomy: impact on continence. J Endourol. 2009 Sep;23(9):1443-50. doi: 10.1089/end.2009.0411. PMID 19698020
- [Background] Finley DS, Chang A, Morales B, Osann K, Skarecky D, Ahlering T. Impact of regional hypothermia on urinary continence and potency after robot-assisted radical prostatectomy. J Endourol. 2010 Jul;24(7):1111-6. doi: 10.1089/end.2010.0122. PMID 20624082
- [Background] Liss MA, Skarecky D, Morales B, Ahlering TE. The application of regional hypothermia using transrectal cooling during radical prostatectomy: mitigation of surgical inflammatory damage to preserve continence. J Endourol. 2012 Dec;26(12):1553-7. doi: 10.1089/end.2012.0345. Epub 2012 Nov 15. PMID 23153199
- See also: Dr. Thomas E. Ahlering, UCI Medical Center — http://www.ucirvinehealth.org/find-a-doctor/a/thomas-ahlering/